CLINICAL TRIAL: NCT02153762
Title: Assessment of Application Order When Utilizing Locoid Lotion and Hylatopic Plus Cream in the Treatment of Atopic Dermatitis
Brief Title: Treatment of Atopic Dermatitis With Different Orders of Application of Locoid Lotion and Hylatopic Plus Cream
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GCO 12-1932
Record Dates: First submitted 2014-05-27; First posted 2014-06-03 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; AD
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Right side (Experimental): Patients were randomized to apply Locoid Lipocream on the right side of the target lesion followed by Hylatopic Plus lotion on the left side of the target lesion with the reverse order on the other side.
  Interventions: Drug: Locoid Lipocream; Drug: Hylatopic Plus
- Left first (Active Comparator): Patients were randomized to apply Locoid Lipocream on the left side of the target lesion followed by Hylatopic Plus lotion on the right side of the target lesion with the reverse order on the other side.
  Interventions: Drug: Locoid Lipocream; Drug: Hylatopic Plus

INTERVENTIONS:
Drug: Locoid Lipocream — Patients were randomized to apply Locoid Lipocream followed by Hylatopic Plus lotion on either the right or left side target lesion with the reverse order on the other side.
  Other Names: Topical skin barrier repair therapies (BRT)
Drug: Hylatopic Plus — Patients were randomized to apply Locoid Lipocream followed by Hylatopic Plus lotion on either the right or left side target lesion with the reverse order on the other side.
  Other Names: Topical skin barrier repair therapies (BRT)

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability, as well as effectiveness, with regards to the order of application for Locoid Lipocream and Hylatopic Plus cream in patients with atopic dermatitis (AD), which is a type of skin rash.Topical skin barrier repair therapies (BRT) that are plain moisturizing creams/lotions with added lipids (fats/oils), such as Hylatopic Plus cream, have emerged as an effective addition to the the treatment of atopic dermatitis. BRTs are often used along with topical steroids (medicated creams), such as Locoid lotion, on skin with AD, and as a monotherapy (single treatment) on both non-diseased and diseased skin. Since BRTs help to restore components of skin that are absent in skin with AD, it is believed that long-term BRT use may reduce further development of further AD. This is an open-label, single site study.

ELIGIBILITY:
Inclusion Criteria:

* subjects of at least 3 months of age.
* clinical diagnosis of stable mild to moderate AD using the Hanifin and Rajka criteria for diagnosing AD
* AD lesions of similar size and severity of bilateral anatomic location
* a SPGA score of 2 or 3 and at least 10% BSA involvement at baseline
* in good health, without evidence of disease process(es) that would present patient safety concerns or confounding factors for assessment of study objectives
* able and willing to understand and sign an informed consent (or if applicable parent or legal guardian sign an informed consent),
* able and willing to agree to requirements and restrictions of the study
* Subjects who are willing to discontinue all systemic corticosteroids, immunomodulators, ultra violet light therapy or other medication (investigational or otherwise) that may have an effect on atopic dermatitis disease progression for 30 days prior to the baseline measurement.
* Subjects on a stable maintenance therapy (at least 30 days of use prior to baseline) of antihistamines and/or nasal spray containing corticosteroids for the treatment of bronchial asthma or allergic rhinitis, and antibiotics for the treatment of acne will be allowed.
* Subjects who are willing to discontinue use of topical treatments for AD including, but not limited to, corticosteroids, immunomodulators, vitamin D treatments, retinoids, topical antihistamines for at least 14 days prior to baseline
* Subjects who are willing to discontinue use of oral antibiotic therapy for at least 7 days prior to baseline, unless prescribed for acne treatment as previously described
* Subjects with no known allergy to any of the study product ingredients
* Women of childbearing potential must be willing to use a form of birth control during the study. For the purpose of this study, the following are considered acceptable methods of birth control: oral contraceptives, Norplant, Depo-Provera, double barrier methods (e.g., condom and spermicide) and abstinence.

Exclusion Criteria:

* immunocompromised patients, or subjects with extensive disease that could not reasonably be controlled with topical therapy
* history or evidence of other conditions that would interfere with the evaluation of the study medication
* subjects desiring excessive or prolonged exposure to UV light (e.g. sunlight/tanning beds) during the study
* Use of topical medications for AD or any other medical condition.
* Subjects currently involved in another clinical research study.
* Subjects, who are pregnant, breast feeding or planning a pregnancy.
* Subjects with clinically significant unstable medical or mental disorders.
* Subjects who are unwilling or unable to comply with the requirements of the protocol.

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Treatment Success at Day 29 | baseline and Day 29
  Treatment Success defined as Clear or Almost Clear (0 or 1) on the 5 point static physician global assessment of psoriasis (SPGA) scale at day 29, evaluating non-inferiority of one group compared to the other using the lower limit of the confidence interval for the difference in success proportions, as compared to baseline.

SECONDARY OUTCOMES:
Change from Baseline SPGA scale at Day 29 | baseline and Day 29
  2 point reduction of SPGA at day 29 as compared to baseline. The sPGA is a physician's global assessment of the participant's psoriasis based on severity of induration, scaling, and erythema. The sPGA of psoriasis comprises a 6-point scale ranging from 0 (clear) to 5 with increasing severity.
Change from Baseline Pruritus at Day 29 | baseline and Day 29
  Change from baseline pruritus at day 29

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Zeichner, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States